CLINICAL TRIAL: NCT06999109
Title: Teams Engaged in Accessible Mental Health Interventions for Lupus Erythematosus and Dermatomyositis Stress
Acronym: TEAM-LEADS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00118057
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Lupus; Dermatomyositis, Juvenile; Dermatomyositis; Lupus Erythematosus; Lupus Erythematosus, Systemic; Lupus or SLE
Keywords: Stress; Depression; Anxiety; Lupus; Dermatomyositis; Pediatric Rheumatology; Physical Activity; Diet Quality; Sleep; Cardiovascular Health; Health Behaviors; Remote Intervention; Online Intervention; Co-Design; Intervention Refinement
MeSH Terms: conditions — Dermatomyositis; Lupus Erythematosus, Systemic; Depression; Anxiety Disorders; Motor Activity; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TEAM-LEADS intervention arm (Experimental)
  Interventions: Behavioral: TEAM-LEADS

INTERVENTIONS:
Behavioral: TEAM-LEADS — TEAM-LEADS will be an online, self-administered intervention for stress reduction and cardiovascular health behavior promotion in adolescents and young adults with juvenile-onset systemic lupus erythematosus and dermatomyositis

SUMMARY:
The objectives of this study are to determine if the 'Teams Engaged in Accessible Mental Health Interventions for Lupus Erythematosus and Dermatomyositis Stress' (TEAM-LEADS) intervention is feasible and acceptable to adolescents and young adults with lupus and dermatomyositis and whether it can help reduce stress and promote cardiovascular health behaviors in these individuals.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of juvenile-onset systemic lupus erythematosus (JSLE) or dermatomyositis (JDM)
* Age 12-22 years old at time of enrollment

Exclusion Criteria:

* Inability to complete surveys/interviews reliably
* Lack of access to internet-enabled device;
* Non-JSLE/JDM diagnosis
* History of myocardial infarction or cerebrovascular accident
* Evidence of severe emotional distress defined as any of the following at time of screening: a) Patient Health Questionnaire for Adolescents (PHQ9A) score ≥ 15 indicating severe depression; b) PHQ9A suicidality item score > 0 indicating presence of any suicidal ideation; c) any other evidence noted of severe emotional distress per PI's judgment.

Ages: 12 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2027-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in Patient-Reported Outcome Measures Information System (PROMIS) Pediatric Psychological Stress Experiences (version 1.0 Short Form 8a) T-scores | From T1 (baseline visit, day 0) to T3 (Day 84)
  T-scores range from 37 to 81.8. Higher T-scores indicate greater psychological stress (i.e. worse outcome).

SECONDARY OUTCOMES:
Change in Cardiovascular Health Behaviors Score | From T1 (baseline visit, day 0) to T3 (Day 84)
  Cardiovascular Health Behaviors Score is a composite of individual measures of diet quality, physical activity, and sleep duration. Scores range 0 to 100. Higher scores indicate better outcomes (i.e., greater presence of cardiovascular health behaviors) with scores = 100 indicating ideal diet quality, physical activity, and sleep duration.

CONTACTS AND LOCATIONS:
Overall Officials: Kaveh Ardalan, MD, MS, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Study protocols, data collection instruments, data dictionaries, and statistical analysis plans will be deposited in Vivli repository via Duke University's institutional license.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be made available at time of publication or the end of the performance period (whichever comes first). At a minimum, Vivli will make data available for researchers for 10 years, unless they are contractually unable to do so.
Access Criteria: Vivli provide metadata, persistent identifiers (e.g. NCT ID), study search functions, and long-term access. Vivli repository is available to Duke investigators via institutional license and datasets are available via standardized process in which requestors search Vivli platform for the study, request the IPD data package (with requests reviewed per contributor's publicly stated requirements), and then access data in Vivli's secure environment (or download with permission).

REFERENCES:
- [Background] Ardalan K, Lloyd-Jones DM, Schanberg LE. Cardiovascular Health in Pediatric Rheumatologic Diseases. Rheum Dis Clin North Am. 2022 Feb;48(1):157-181. doi: 10.1016/j.rdc.2021.09.006. Epub 2021 Oct 29. PMID 34798945